CLINICAL TRIAL: NCT06854822
Title: Siblings to a Child with Cancer: Psychometric Evaluations of Instruments Assessing Siblings Needs and Pre-loss Grief
Brief Title: Siblings to a Child with Cancer: Needs and Pre-loss Grief
Status: Recruiting | Type: Observational
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Malin Lövgren, Professor, Ersta Sköndal University College
Other Study IDs: 2023-03752-01
Record Dates: First submitted 2025-01-29; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Childhood Cancer; Siblings; Psychosocial Functioning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background and Aim: Siblings to a brother or sister with cancer have reported difficulties dealing with such things as their parents' suffering, loneliness in relation to their own feelings as well as uncertainty regarding their brother's/sister's treatment, prognosis and survival. Siblings also struggle with fear of death and dying, and unresolved grief. Unfortunately, siblings are a forgotten group both in society, within the family, in health care, in school, and in research even if there has been a huge improvement the last 10 years. These children's needs must be identified and handled during the illness trajectory as a way of supporting their challenging situation and prevent avoidable psychological distress. Nevertheless, there exists no validated standardized assessment instrument in Swedish that measure the needs of these children even if it is well known that it is beneficial for emotional and psychological well-being to use assessment instrument. Moreover, no instrument in Swedish exists that identify children with prolonged pre-death grief despite that prolonged grief during illness is associated with psychological distress. This study therefore aim to translate, culturally adapt, and evaluate the psychometric properties of the Swedish version of the Sibling Cancer Needs Instrument (SCNI) and Prolonged Grief Disorder (PG-12) among children and youths who have a brother or sister with cancer.

Material and Methods: Present instruments will be translated and culturally adapted according to the World Health Organization's (WHO) guidelines. After that, the psychometric properties of the Swedish version of SCNI and PG-12 will be examined. The Swedish version of the SCNI and PG-12 will be revised by a group of several experts in psychology, paediatric oncology, and family health, for its face and content validity. In addition, pre-test respondents will include approx. 10 siblings. They will be recruited from one of the six pediatric oncology centers in Sweden, the home care for children at the same hospital, and at the hospice for children and youths in Sweden (Lilla Erstagården) where established collaborations with clinicians exists today with sibling supporters. Information about the study will be given by the researchers who also ask for informed consent. Children aged 15 years and older consent themselves while those between 12-14 years have to have consent from their guardian(s)/parent(s). Pre-test respondents will be administered SCNI and PG-12 and be systematically debriefed. During debriefing, siblings will be asked what they thought the question was asking, whether they could repeat the question in their own words, what came to their mind when they heard a particular phrase or term. They will also be asked to explain how they choose their answer. These questions will be repeated for each item. The answers to these questions should be compared to the respondent's actual responses to the instrument for consistency. Respondents will also be asked about any word they did not understand as well as any word or expression that they found unacceptable or offensive. Finally, when alternative words or expressions exist for one item or expression, the pre-test respondent should be asked to choose which of the alternatives conforms better to their usual language. After that, siblings will be asked to participate in a web-survey. They will be recruited from: 1) the six pediatric oncology centers in Sweden, 2) the hospice for children and youths in Sweden (Lilla Erstagården), and 3) via advertisement on social media, e.g. on Instagram at "Nära Cancer" and the Childhood Cancer Fund. The siblings will also be identified by a sibling supporter at the six pediatric oncology centers and Lilla Erstagården. The sibling supporters will invite the siblings to the study by giving them a web address to a website where they will find information about the study. On the website, the siblings could either go directly to the web-survey (if the sibling is 15 years or older) or register their interest to participate in the web-survey (if the sibling is between 12-14 years). Parents of siblings who register their interest to participate in the web-survey on the website (siblings aged 12-14 years), will be contacted by a researcher via email or phone (depending on how they wish to be contacted), and the parents/guardians and the sibling will be informed about the study, and informed consent will be granted from both guardians/parents. Advertisement on social media will take the siblings or parents/guardians to the same web-page/web-survey as previously described.

Analysis: Descriptive statistics will be used to present demographic data and study variables, including means and standard deviations, medians and quartiles, and frequencies. We will use factor analysis in order to evaluate the fit of the models. A sample size of 200 will be acceptable if the models are not too complex.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-24 years
* Have a brother or sister with childhood cancer
* Swedish speaking siblings

Exclusion Criteria:

-Bereaved siblings

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All siblings that have a brother or sister with cancer 0-17 years.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Psychosocial needs | Through study completion, an average of 1 year
  The Sibling Cancer Need Instrument (SCNI) will be used as primary outcome. SCNI is developed for siblings in the age of 12-24 years. SCNI has 45 items and seven domains: information; practical assistance; "time out" and recreation; feelings; support (friends and other young people); understanding from my family; and sibling relationship. The instrument contains the sentence stem 'I currently need....', and responses use a 4-item response scale where: 1=no need, 2=low need, 3=moderate need, and 4= strong need. The possible range of scores is 45-180, with higher scores indicating more unmet needs.

SECONDARY OUTCOMES:
Pre-grief | Through study completion, an average of 1 year
  Prolonged grief disorder (PG12). PG-12 covers: 1) separation distress, which is characterized by manifestations of longing and yearning, 2) emotional, cognitive, and behavioural symptoms, e.g., diminished sense of self, feeling stunned or shocked by the patient's illness, having trouble accepting it, and feelings of meaninglessness, and 3) social and occupational functioning. A summary score for the symptom items is calculated by totaling each individual item score from 1 (not at all) to 5 (overwhelmingly). Symptom scores can range from 10 to 50. A score of 30 or greater indicates higher levels of PGD.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Lövgren, PhD, Principal Investigator — Marie Cederschiöld University
Locations (1):
- Marie Cederschiöld Unicersity College, Stockholm, Sweden